CLINICAL TRIAL: NCT07331311
Title: Evaluation of Diagnostic Benefit and Feasibility of Using Lung Ultrasound to Diagnose Childhood Pneumonia in Low-resource Settings
Brief Title: Diagnostic Accuracy of Lung Ultrasound for Pneumonia Diagnosis in Children
Acronym: LUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nagasaki University (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Global Health Research and Medical Interventions Institute (GlohMed), Nepal (Unknown)
Responsible Party: Principal Investigator, Suraj BHATTARAI, Research fellow (WISE programme), Nagasaki University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 31322
Record Dates: First submitted 2025-12-16; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Pneumonia; Childhood Pneumonia
Keywords: Lung ultrasound; Point-of-Care test; Point-of-Care Lung Ultrasound
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Intervention Model Description: Lung ultrasound followed by chest X-ray in all enrolled participants as chest imaging investigation
Masking Description: Care provider performing LUS scans are masked of CXR report and clinical information about he participant, other than the case has WHO defined pneumonia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chest imaging (Experimental): Single arm study that evaluates the role of LUS in diagnosing pneumonia in children. All participants receive LUS scans followed by CXR as chest imaging intervention.
  Interventions: Diagnostic Test: LUS as a chest imaging tool

INTERVENTIONS:
Diagnostic Test: LUS as a chest imaging tool — Each study participant receives LUS scan followed by CXR as chest imaging modality. LUS is the diagnostic test under investigation, compared against clinical gold standard (described later).

SUMMARY:
Chest X-ray is historically being used as an imaging standard to aid to the diagnosis of childhood pneumonia, however, the evidence does not support it as a perfect imaging tool. As an alternative to CXR, lung ultrasound (LUS) could be used as the imaging of choice in children and studies have demonstrated its good accuracy to diagnose childhood pneumonia. However, most diagnostic studies have used CXR as a reference standard.

In absence of a 'gold standard' approach, there is a risk that large proportion of children with pneumonia and severe pneumonia could be 'missed' if clinicians relied on LUS only.

This research aims to evaluate the diagnostic benefit of LUS in children compared against 'gold standard' diagnosis which is derived based on the clinical information, imaging and laboratory investigations.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of pneumonia. Pneumonia is suspected in a child meeting the WHO case definition of pneumonia, i.e. cough or difficulty breathing associated with fast breathing and/ or lower chest wall indrawing.

Exclusion Criteria:

* Non-consenting parents.
* Children who are hospitalized for more than 24 hours.
* Children treated for pneumonia at the study site within past 4 weeks.
* Critical patients requiring emergency lifesaving support and parents unable to cooperate to provide consent.

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Pneumonia missed by LUS | From enrolment until day-5 follow up
  Proportion of children with any pneumonia (severe or non-severe) that would be missed by LUS at initial presentation
Pneumonia missed by CXR | From enrolment until day-5 follow up
  Proportion of children with any pneumonia (severe or non-severe) that would be missed by CXR at initial presentation

SECONDARY OUTCOMES:
Diagnostic accuracy of LUS | From enrolment to day-5 follow up
  Sensitivity and specificity of LUS for pneumonia diagnosis in children, compared against 'Gold standard' diagnosis adjudicated by expert paediatrician panel after reviewing all available clinical information about the child during study time frame
Diagnostic accuracy of CXR | From enrolment to day-5 follow up
  Sensitivity and specificity of CXR for pneumonia diagnosis in children, compared against 'Gold standard' diagnosis adjudicated by expert paediatrician panel after reviewing all available clinical information about the child during study time frame

OTHER OUTCOMES:
Proportion of 'missed pneumonia' cases with adverse clinical outcomes | From day of enrolment to day-5 follow up
  List of adverse clinical outcomes and their measures:
  1. 'Clinical worsening' - defined as change from non-severe pneumonia to severe pneumonia status;
  2. 'Development of pulmonary complications' - defined as development of pleural effusion, empyema, pneumatocele, TB or respiratory failure/ARDS requiring ventilator support for the current episode of illness;
  3. 'ICU admission' - defined as requiring ICU care for current episode of illness;
  4. 'Revisit or readmission' - defined as unscheduled ER visit and/ or readmission within 4 weeks of initial visit for current episode of illness;
  5. 'Prolonged hospitalisation' - defined as hospitalisation for more than 5 days;
  6. 'Mortality' - if the child died due to current episode of illness

CONTACTS AND LOCATIONS:
Overall Officials: Suraj Bhattarai, MBBS, MSc, DTM&H, Principal Investigator — London School of Hygiene and Tropical Medicine/ Nagasaki University School of Tropical Medicine and Global Health
Locations (1):
- Siddhi Memorial Hospital, Bhaktapur, Bagmati, Nepal